CLINICAL TRIAL: NCT04862325
Title: SOPHIE: Surgery in Ovarian Cancer With PreHabilitation In ERAS: Prospective Multicentre Study
Brief Title: SOPHIE Trial: Surgery in Ovarian Cancer With PreHabilitation In ERAS
Acronym: SOPHIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Berta Diaz-Feijoo, Study Director, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HCB/2020/0317
Record Dates: First submitted 2021-04-12; First posted 2021-04-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Advanced Ovarian Cancer
Keywords: Prehabilitation; Advanced ovarian cancer; cytoreductive surgery; postoperative complications; exercise training; nutrition; physical activity; mindfulness meditation
MeSH Terms: conditions — Postoperative Complications; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Control group will follow the standard preoperative measures "Enhanced Recovery After Surgery" (ERAS®) established in the protocols of our hospital. Standard preoperative measures: recommendation of nutritional and physical activity and advice to stop smoking and reduce alcohol intake; optimization of preoperative pathologies including anaemia. An information document on ERAS® measures in our center will be attached to all of them.
- Multimodal prehabilitation (Experimental): Patients following the standard preoperative policies of our institution and the multimodal prehabilitation program
  Interventions: Other: Multimodal Prehabilitation

INTERVENTIONS:
Other: Multimodal Prehabilitation — 1. High-intensity endurance exercise training program and physical activity promotion remotely controlled with ICT (information and communications technologies).
  2. Nutritional counselling to achieve protein intake of 1.5-1.8 g/kg and whey protein supplements.
  3. Psychological intervention including motivational interview, mindfulness meditation and cognitive behavioral therapy
  Arms: Multimodal prehabilitation

SUMMARY:
The treatment of choice in advanced ovarian cancer is a cytoreductive surgery combined with chemotherapeutic treatment. This complex and aggressive surgery is associated with high postoperative complication rates that may result in a strong negative impact on the clinical results due to the delay with the start of adjuvant chemotherapy as well as the costs from the surgical process. Multimodal prehabilitation has emerged as an innovative intervention that focuses on optimizing physiological and psychological resilience to withstand the upcoming stress of surgery. It has been shown to reduce postoperative complications in major abdominal surgery, but has not been assessed yet in abdominal onco-gynecological surgery.

DETAILED DESCRIPTION:
Main objective: To determine the efficacy of multimodal prehabilitation in decreasing postoperative complications in patients undergoing gynecological cancer surgery of high complexity by laparotomy (primary cytoreductive surgery, interval surgery and secondary cytoreductive surgery in advanced ovarian cancer).

Design: Multicenter randomized controlled clinical trial. Subjects: 146 patients: 73 in the intervention group and 73 in the control group.

Intervention group: PreHAB intervention consists on:

1. High-intensity endurance exercise training program and physical activity promotion remotely controlled with ICT (information and communications technologies).
2. Nutritional counselling to achieve protein intake of 1.5-1.8 g/kg and whey protein supplements.
3. Psychological coping. Control group will receive standard preoperative care. Both groups will receive perioperative care in accordance with the enhanced recovery after surgery (ERAS) guidelines.

Measures: Aerobic capacity (incremental stress test), physical activity, operative complications and hospital length and associated costs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced ovarian cancer subject to primary debulking surgery or interval surgery after 3-4 cycles of chemotherapy or secondary and / or tertiary debulking surgery .
2. Patients with Eastern Cooperative Oncology Group (ECOG) performance status 2-0.
3. Adherence of at least 75 % of the program or minimum of 6 sessions.

Exclusion Criteria:

1. Surgery without a minimum of 3 weeks of prehabilitation time.
2. Unstable respiratory or heart disease.
3. Locomotor or cognitive limitations that makes not feasible the adherence to the program.
4. Refusal of the patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications | 30 days
  Any deviation from the normal postoperative course and according its severity to the Clavien-Dindo classification, will be considered a complication.
  A comprehensive complication index (CCI) scale will be used which assigns a value to each Clavein-Dindo level so a weighted average of the severity of complications can be calculated not only in a qualitatively way, but also numerically.

SECONDARY OUTCOMES:
Hospital and ICU (intensive care unit) length of stay | postoperative 30 days
Compliance to the ERAS program. | postoperative 30 days
  Percentage of items of ERAS program that were completed. Key aspects of this protocol include prevention of prolonged fasting allowing oral intake of clear fluids up to 2 hours before induction of anaesthesia, carbohydrate loading, avoidance of mechanical bowel preparation except if a bowel resection is scheduled, thromboprophylaxis; pre-, intra-, and post-operative euvolemia via goal directed fluid therapy, maintenance of normothermia, intraoperative and postoperative opioid-sparing multi-modal analgesia, avoidance the use of surgical drains, early removal of the urine catheter, and an emphasis on early ambulation and feeding.
Interval of days between surgery and the start of chemotherapy | From date of surgery up to 6 months
Preoperative and postoperative aerobic capacity | baseline, 1 and 3 month post intervention
  Maximum production of carbon dioxide in ml/min during high intensity cardiopulmonar exercise.
Cost-effectiveness | Baseline up to 30 days after surgery
  Cost of treatment in the hospital in Euros including prehabilitation and postoperative recovery.
Health Related Quality of Life assesed by EORTC QLC-C30 | Baseline and 1 month postoperative
Incidence of cognitive deficit | Baseline and 1 month postoperative
  Cognitive assessment based on validated neuropsychological test: T @ M (; Digits WAIS III (Wechsler Adult Intelligence Scale-Third Edition)
Overall and disease-free survival of the study groups | 5 years
Nutritional status | Baseline and 1 month postoperative
  GLIM (includes hand-grip)

CONTACTS AND LOCATIONS:
Overall Officials: Berta Diaz-Feijoo, MD PHD, Principal Investigator — Hospital Clinic of Barcelona; M Jose Arguis, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Biomedical Research Institute la Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Derived] Diaz-Feijoo B, Agusti N, Sebio R, Siso M, Carreras-Dieguez N, Domingo S, Diaz-Cambronero O, Torne A, Martinez-Palli G, Arguis MJ. A multimodal prehabilitation program for the reduction of post-operative complications after surgery in advanced ovarian cancer under an ERAS pathway: a randomized multicenter trial (SOPHIE). Int J Gynecol Cancer. 2022 Nov 7;32(11):1463-1468. doi: 10.1136/ijgc-2022-003652. PMID 35793862